CLINICAL TRIAL: NCT01639066
Title: A Multicenter Randomized Controlled Open-label Trial of Tenofovir Plus Entecavir Combination vs. Tenofovir Monotherapy in Chronic Hepatitis B Patients With Genotypic Resistance to Adefovir and Partial Virologic Response to Ongoing Treatment
Brief Title: Tenofovir Plus Entecavir vs. Tenofovir in Adefovir-Resistant Chronic Hepatitis B
Acronym: IN-US-0205
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Konkuk University Medical Center (Other); Korea University Guro Hospital (Other); Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Young-Suk Lim, Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC2012-1208
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Chronic Viral Hepatitis B Without Delta-agent
Keywords: Resistance of Adefovir
MeSH Terms: interventions — Tenofovir; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tenofovir plus Entecavir combination (Experimental): Tenofovir 300 mg/day orally and Entecavir 1 mg/day orally
  Interventions: Drug: Tenofovir; Drug: Entecavir
- Tenofovir monotherapy (Active Comparator): Tenofovir 300 mg/day orally
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir — Tenofovir 300mg daily Oral
  Other Names: Viread
  Arms: Tenofovir plus Entecavir combination
Drug: Entecavir — Entecavir 1 mg daily Oral
  Other Names: Baraclude
  Arms: Tenofovir plus Entecavir combination
Drug: Tenofovir — Tenofovir 300mg daily Oral
  Other Names: Viread
  Arms: Tenofovir monotherapy

SUMMARY:
With the availability of potent nucloes(t)ide analogues (NA), such as tenofovir disoproxil fumarate (TDF) and entecavir (ETV), suppression of serum HBV DNA to undetectable levels by polymerase chain reaction (PCR) assays became achievable in most NA treatment-naïve patients. Until recently, however, many patients commenced antiviral treatment with inferior NAs prior to the availability of TDF or ETV, such as lamivudine (LAM) or adefovir (ADV) which has a low genetic barrier to resistance.

For patients who developed genotypic resistance against ADV, the efficacy of TDF monotherapy is controversial. In recent studies, TDF monotherapy produced significant suppression of HBV replication. However, only half of patients with initial ADV resistance achieved an undetectable viral load (<15 IU/ml) with 48 weeks of therapy.

On the other hand, there was a retrospective cohort study reporting that, with the combination of TDF and ETV, most of patients became HBV DNA undetectable after median 6 months of treatment. Probability of reaching complete HBV DNA suppression was not decreased in patients with ADV or ETV resistance.

Together, these observations indicate that there is a controversy about the efficacy of TDF monotherapy in patients with genotypic resistance to ADV.

Thus, in this clinical trial, the investigators will clarify whether tenofovir monotherapy is effective in inducing complete virologic response compared with tenofovir plus entecavir in CHB patients with genotypic resistance to ADV and partial virologic response to ongoing treatment.

DETAILED DESCRIPTION:
A multi-center randomized active-controlled open-label trial

* Patients will be randomly assigned 1:1 to receive tenofovir (300 mg/day) or tenofovir (300 mg/day) plus entecavir (1 mg/day) for 48 weeks.
* Because over 98% of Korean patients with CHB have HBV genotype C, HBV genotype will not be determined or be regarded as a stratification factor.
* Patients' treatment information before randomization will be retrospectively collected.(DNA change, HBeAg status, HBsAg titre, ALT, and treatment duration. etc)
* Patients will be screened within 4 weeks before randomization to determine study eligibility.

ELIGIBILITY:
Inclusion Criteria: All of below

* Compensated liver disease (Child-Pugh class A)
* HBsAg positive at least 6 months or more
* HBeAg positive or negative
* Confirmation of ADV resistance mutation at any time before screening (rtA181V or rtA181T or rtN236T)
* Serum HBV DNA ≥ 60 IU/mL despite continued preceding oral antiviral treatment (Serum HBV DNA should be determined by the PCR assay at the local laboratory at screening for this study)
* Patient is ambulatory.
* Patient is willing and able to comply with the study drug regimen and all other study requirements.
* The patient is willing and able to provide written informed consent to participate in the study.

Exclusion Criteria: Any of below

* Patient previously received TDF for more than 1 week
* Patient has a history of hepatocellular carcinoma (HCC) or findings suggestive of possible HCC, such as suspicious foci on imaging studies. In patients with such findings, HCC should be ruled-out prior to randomizing the patient for the present study.
* Patient has received interferon or other immunomodulatory treatment for HBV infection in the 12 months before screening for this study.
* Patient has concomitant other chronic viral infection (HCV or HIV)
* Patient has evidence of renal insufficiency defined as serum creatinine > 1.5 mg/dL
* Patient has medical condition that requires concurrent use of systemic prednisolone or other immunosuppressive agent (including chemotherapeutic agent)
* Patient is currently abusing alcohol (more than 40 g/day) or illicit drugs, or has a history of alcohol abuse or illicit substance abuse within the preceding two years.
* Patient is pregnant or breastfeeding or willing to be pregnant
* Patient has one or more additional known primary or secondary causes of liver disease, other than hepatitis B (e.g., alcoholism, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's Disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease, etc.).
* A history of treated malignancy (other than hepatocellular carcinoma) is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding three years.
* Clinical signs of decompensated liver disease as indicated by any one of the following:

  1. serum bilirubin > 3 mg/dL
  2. prothrombin time > 6 seconds prolonged or INR >1.5
  3. serum albumin < 2.8 g/dL
  4. History of ascites, variceal hemorrhage, or hepatic encephalopathy
  5. Child-Pugh score ≥7

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-09-25 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete virologic response | at week 48 of treatment
  The proportion of patients who achieve complete virologic response (serum HBV DNA concentrations below 15 IU/mL)

SECONDARY OUTCOMES:
Changes in serum HBV DNA levels | at week 48, 96, 144, and 240 of treatment
  Changes in serum HBV DNA levels during 48 weeks of treatment
Proportion of patients with normal ALT | at week 48, 96, 144, and 240 of treatment
Proportion of patients with HBe-Ag loss or seroconversion | at week 48, 96, 144, and 240 of treatment
Proportion of patients with resistance mutations to Adefovir, Entecavir, or Tenofovir | at week 48, 96, 144, and 240 of treatment
  The proportion of patients with resistance mutations to Adefovir, Entecavir, or Tenofovir at week 48
Proportion of patients with virologic breakthrough | at week 48, 96, 144, and 240 of treatment
  Virologic breakthrough is defined as the increase in serum HBV DNA by >1 log10 (10-fold) above nadir after achieving virologic response as determined by at least 2 consecutive measurements of at least 2 weeks apart, during continued treatment
Proportion of patients with complete virologic response | at week 48, 96, 144, and 240 of treatment
  The proportion of patients who achieve complete virologic response (serum HBV DNA concentrations below 15 IU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Young-Suk Lim, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Lim YS, Yoo BC, Byun KS, Kwon SY, Kim YJ, An J, Lee HC, Lee YS. Tenofovir monotherapy versus tenofovir and entecavir combination therapy in adefovir-resistant chronic hepatitis B patients with multiple drug failure: results of a randomised trial. Gut. 2016 Jun;65(6):1042-51. doi: 10.1136/gutjnl-2014-308435. Epub 2015 Mar 23. PMID 25800784
- [Derived] Lim YS, Gwak GY, Choi J, Lee YS, Byun KS, Kim YJ, Yoo BC, Kwon SY, Lee HC. Monotherapy with tenofovir disoproxil fumarate for adefovir-resistant vs. entecavir-resistant chronic hepatitis B: A 5-year clinical trial. J Hepatol. 2019 Jul;71(1):35-44. doi: 10.1016/j.jhep.2019.02.021. Epub 2019 Mar 13. PMID 30876946
- Available data/document: pubmed: 25800784 — http://www.ncbi.nlm.nih.gov/pubmed/25800784 — Publication for the primary study results